CLINICAL TRIAL: NCT05565599
Title: An Early Feasibility Study Evaluating the Safety and Efficacy of the Laminar Left Atrial Appendage Closure System in Subjects With Non-Valvular Atrial Fibrillation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAM202404; CL-0043 (Other: Biosense Webster, Inc.)
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Non-valvular Atrial Fibrillation
MeSH Terms: interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Closure of the left atrial appendage with the Laminar Left Atrial Appendage Closure system.
  Interventions: Device: Left Atrial Appendage Closure

INTERVENTIONS:
Device: Left Atrial Appendage Closure — Closure of the left atrial appendage with the Laminar Left Atrial Appendage Closure System.

SUMMARY:
This is an early feasibility study is to evaluate the safety and effectiveness of the Laminar Left Atrial Appendage Closure System to treat patients with non-valvular atrial fibrillation that cannot take, or a have a reason to seek an alternative, to anticoagulant medications.

DETAILED DESCRIPTION:
Left atrial appendage closure (LAAC) is an approved therapy for stroke prevention in atrial fibrillation patients who are recommended for chronic oral anticoagulation therapy (OAC), but are non-eligible or have an appropriate rationale to seek a non-pharmacologic alternative to chronic oral anticoagulants in accordance with evidence-based decision-making criteria and current scientific guidelines.

The objective of this study is to evaluate the safety and effectiveness of the Laminar Left Atrial Appendage Closure System to treat patients with non-valvular atrial fibrillation who are deemed appropriate for LAAC to reduce the risk of stroke and systemic embolism.

Patients will be followed for 5 years after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Documented non-valvular AF, defined as AF (paroxysmal, persistent, or permanent) in the absence of moderate-to-severe mitral stenosis or a mechanical heart valve.
2. Subject ≥18 years old.
3. CHA2DS2-VASc score ≥ 2 in men and ≥ 3 in women.
4. Subject is recommended for chronic oral anticoagulation therapy (OAC) but is not eligible or has an appropriate rationale to seek a non-pharmacologic alternative to chronic OAC.
5. Subject deemed appropriate for LAA closure by the Site Heart Team using an evidenced based decision-making tool.
6. Subject eligible for the protocol-specified post-procedural antithrombotic regimen.
7. Subject or Legally Authorized Representative informed of the nature of the study, is willing and able to comply with the protocol, and has provided written informed consent per Institutional Review Board (IRB) requirements.

Exclusion Criteria:

1. Single episode, transient, or reversible AF (e.g., secondary thyroid disorders, acute alcohol intoxication, trauma, recent major surgical procedures).
2. Stroke or transient ischemic attack within 90 days before the index procedure.
3. Myocardial infarction or unstable angina within 90 days before the index procedure.
4. Renal insufficiency, defined as estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2, or dialysis at the time of screening.
5. Active infection with bacteremia.
6. Confirmed COVID-19 infection within 10 days before the index procedure. Coexisting Cardiovascular Disease
7. Cardiac tumor
8. History of mitral valve or other severe cardiac valvular disease requiring intervention or presence of prosthetic mechanical valve.
9. Medical condition (other than AF) that mandates chronic oral anticoagulation (e.g., history of unprovoked deep vein thrombosis or pulmonary embolism, or mechanical heart valve).
10. Severe heart failure (New York Heart Association Class IV).
11. Symptomatic carotid artery disease (>50% diameter reduction with prior ipsilateral stroke or TIA) or asymptomatic carotid artery disease (diameter reduction of >70%).

    Previous or Planned Interventions
12. Previous AF ablation procedure in the 90 days before the index procedure date or need for AF ablation to be performed in less than 90 days after the index procedure.
13. Recent (within 30 days before the index procedure) or planned (within 60 days after the index procedure) cardiac or non-cardiac interventional or surgical procedure.
14. Intracardiac thrombus or dense spontaneous echo contrast visualized by TEE within 2 days before the index procedure.
15. Left ventricular ejection fraction (LVEF) <30%.
16. Circumferential pericardial effusion >10 mm or symptomatic pericardial effusion, signs or symptoms of acute or chronic pericarditis, or evidence of tamponade physiology.
17. Complex atheroma with mobile plaque of the aorta.
18. Interatrial communication, atrial septal defect, or patent foramen ovale that warrants closure.
19. Vascular access precluding delivery of implant with catheter-based system
20. Presence of inferior vena cava (IVC) filter that would interfere with Laminar sheath insertion.
21. Subject unable to undergo general anesthesia.
22. Subject with condition which precludes adequate transesophageal echocardiographic (TEE) assessment.
23. Known allergy, hypersensitivity or contraindication to aspirin, heparin, or device materials (e.g., nickel, titanium).
24. Contrast sensitivity that cannot be adequately pre-medicated.
25. Bleeding diathesis or coagulopathy
26. Thrombocytopenia (platelet count <75,000 cells/mm3), thrombocytosis (>700,000 cells/mm3), or leukopenia (white blood cell count <3,000 cells/mm3).
27. Pregnant or nursing and those who plan pregnancy in the period up to 1 year following the index procedure. Subjects of childbearing potential must have a negative pregnancy test (per site standard test) within 7 days before index procedure.
28. Known other medical illness or known history of substance abuse that may cause non-compliance with the protocol or protocol-specified medication regimen, confound the data interpretation, or is associated with a life expectancy of less than 1 year.
29. Current participation in another investigational drug or device study that in the opinion of the investigator could confound the data interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Composite Adverse Events | 45 days
  Composite rate of all-cause mortality, stroke, systemic embolism, life threatening or major bleeding (BARC Type 3 or 5), pericardial effusion requiring drainage, device embolization, and device- or procedure-related events requiring open cardiac surgery or major endovascular intervention.
Composite Adverse Events | 12 months
  Composite rate of all-cause mortality, stroke, systemic embolism, life threatening or major bleeding (BARC Type 3 or 5), pericardial effusion requiring drainage, device embolization, and device- or procedure-related events requiring open cardiac surgery or major endovascular intervention.
LAA Closure Rate | 45 days
  Rate of LAA closure defined by peri-device flow ≤ 3mm in width per TEE evaluated by independent core laboratory.
LAA Closure Rate | 12 months
  Rate of LAA closure defined by peri-device flow ≤ 3mm in width per TEE evaluated by independent core laboratory.
LAA Closure Rate | 45 days
  Rate of LAA closure per CCTA evaluated by independent core laboratory. Contrast patency defined as LAA density ≥100 HU or ≥25% of that of the left atrium.
Composite of Ischemic Stroke or System Embolism | 12 months
  Composite of ischemic stroke or systemic embolism.

SECONDARY OUTCOMES:
Device-Related Thrombus | 45 days
  Rate of device-related thrombus (DRT) per CCTA evaluated by independent core laboratory.
Device-Related Thrombus | 12 months
  Rate of DRT per TEE evaluated by independent core laboratory.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Tucson Medical Center, Tucson, Arizona
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - Scripps Health, La Jolla, California
  - UC Davis Medical Center, Sacramento, California
  - Los Robles Hospital & Medical Center, Thousand Oaks, California
  - The Mount Sinai Hospital, New York, New York
  - Columbia U. Medical Center / NY Presbyterian Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No